CLINICAL TRIAL: NCT03536169
Title: Utilization of Anti-reflux Treatment and Course of Illness Leading to Reoperation After Anti-reflux Surgery in a National Population-based Cohort
Brief Title: Utilization of Anti-reflux Treatment and Course of Illness Leading to Reoperation
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense Patient Data Explorative Network (Other); Kolding Sygehus (Other)
Responsible Party: Principal Investigator, Jonas Sanberg Jensen, MD, Ph.d.-student, University of Southern Denmark
Other Study IDs: JSJ_OP446
Record Dates: First submitted 2018-05-09; First posted 2018-05-24 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: GERD; Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate course of illness leading to reoperation after primary anti-reflux surgery and investigate the utilization of anti-reflux treatment, both medical and surgical, in the period 2000-2017

DETAILED DESCRIPTION:
Aim The purpose of this study is to investigate course of illness leading to reoperation after primary anti-reflux surgery and investigate the utilization of anti-reflux treatment, both medical and surgical, in the period 2000-2017

Methods The study is a two-part register-based cohort study based on data from The National Patient Registry, The Civic Registry and Danish Anaesthesia Database in the period 1996-2017. The two individual parts of the study concerns the same population.

The population is defined as all adult Danish patients undergoing anti-reflux surgery (Nomesco: KJBC00, KJBC01, KJBC02, KJBW96, KJBW97) from 2000-2017 identified from The National Patient Register.

Age, sex, Charlson Comorbidity Index at date of surgery and length of stay in relation to any surgery and any surgical or endoscopic procedure performed after anti-reflux surgery (including diagnosis 30 days postoperatively to establish possible morbidity) are derived from the National Patient Registry.

ASA-score, weight, height, use of alcohol or tobacco and priority of any surgery (emergency or planned) during the study period are retrieved from The Danish Anaesthesia Database. From the Civic Register, data on mortality in the study period are retrieved.

Information on the use of pharmacological treatment for gastroesophageal reflux disease on population level is retrieved from MEDSTAT and data on population size on population level are retrieved from Statistics Denmark.

Statistical analysis

1. Course of illness leading to reoperative anti-reflux surgery Data will be analyzed using STATA15. Descriptive analysis of age, sex, comorbidity (Charlson Comorbidity Index, ASA-score, BMI, alcohol/tobacco use), complications to surgery, rate of endoscopic dilation and mortality comparing patients with only primary anti-reflux surgery and patients with reoperation during the study period, will be performed using Student's t-test, Chi2-test and Mann-Whitney-U test.

   Logistic regression will be performed with reoperation (laparoscopic, open or other) as primary outcome and age, sex, comorbidity (Charlson Comorbidity Index, ASA-score, BMI, alcohol/tobacco use), complications to surgery and endoscopic or surgical procedure during study period as independent variables. If the number of patients is sufficient, subanalysis will be performed with emergency reoperation as dependent variable/outcome.

   Secondary analysis will be performed using Cox-regression investigating time to reoperation with age, sex, comorbidity (Charlson Comorbidity Index, ASA-score, BMI, alcohol/tobacco use), complications to surgery and endoscopic or surgical procedure during study period as independent variables.
2. Utilization of treatment of gastroesophageal reflux disease. The rate of anti-reflux surgery per 100.000 inhabitants for each year during the study period will be calculated using census data from Statistics Denmark. From MEDSAT the rate of use of pharmacological anti-reflux treatment per 100.000 inhabitants will be calculated using abovementioned census-data. Trends in the utilization of surgery are investigated with trend-analysis in the form of Poisson-regression alternatively negative binominal regression.

ELIGIBILITY:
Inclusion Criteria:

* All adult Danish patients undergoing anti-reflux surgery (Nomesco: KJBC00, KJBC01, KJBC02, KJBW96, KJBW97) from 2000-2017 identified from The National Patient Register.

Exclusion Criteria:

* Any diagnosis of gastrointestinal cancer during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is defined as all adult Danish patients undergoing anti-reflux surgery (Nomesco: KJBC00, KJBC01, KJBC02, KJBW96, KJBW97) from 2000-2017 identified from The National Patient Register.
Sampling Method: Non-Probability Sample
Enrollment: 3717 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Reoperation | 2000-2017 (Maximum of 17 years follow-up, minimum of 1 year)
  Any reoperative anti-reflux surgery
Rate of anti-reflux surgery | 2000-2017
  Based on Danish census-data
Rate of pharmacological anti-reflux treatment | 2000-2017
  Based on Danish census-data

SECONDARY OUTCOMES:
Emergency reoperative anti-reflux surgery | 2000-2017(Maximum of 17 years follow-up, minimum of 1 year)
  Rate of reoperative surgery performed as emergency procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jonas S Jensen, MD, Principal Investigator — Department of Surgery, Kolding Hospital
Locations (1):
- Department of Surgery, Kolding Hospital, Kolding, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual patient data are by Danish law no allowed to be shared without specific authorization prior to study initiation.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/69/NCT03536169/Prot_SAP_000.pdf